CLINICAL TRIAL: NCT00916188
Title: Effects of Black Tea Consumption on Oxidative Stress, Serum Lipid Profile and Insulin Sensitivity in Patients With Type 2 Diabetes
Brief Title: Effects of Black Tea on Type 2 Diabetes
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: National Nutrition and Food Technology Institute (Other)
Responsible Party: Tirang reza Neyestani, National Nutrition and Food Technology Institute
Allocation: Randomized | Model: Parallel | Masking: None
Other Study IDs: P/25/47/4564
Record Dates: First submitted 2009-06-08; First posted 2009-06-09 (Estimated); Last update posted 2010-07-27 (Estimated); Status verified 2009-06

CONDITIONS: Type 2 Diabetes Mellitus
Keywords: Black Tea; Oxidative Stress; Blood Lipids; Insulin Sensitivity
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Insulin Resistance | interventions — Tea

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Black Tea-Four Doses (Experimental): One, 2, 3 and 4 cups (150 ml/cup) of Black tea/day for week 1, 2, 3, and 4, respectively.
  Interventions: Dietary Supplement: Black Tea Extract
- Black Tea-One Dose (Active Comparator): One cup (150 ml) of Black tea/day during study.
  Interventions: Dietary Supplement: Black Tea Extract

INTERVENTIONS:
Dietary Supplement: Black Tea Extract — Amount/dose depends on Arm assignment.
  Other Names: BTE

SUMMARY:
The primary objective of this study is to evaluate the efficacy of different doses of black tea (150, 300, 450, 600 ml) in the test group compared to 150 ml in the control group, in improving oxidative stress, lipid profiles and insulin sensitivity.

DETAILED DESCRIPTION:
A total of 45 patients of known T2DM (16 males and 29 females) were introduced into the controlled clinical trial and randomly assigned to either test (57.0 ± 7.9 yrs, n=23) or control (55.4 •± 8.3 yrs, n=22) group. Patients in control group were instructed to have only one cup (150 ml) of black tea/day, as a 2.5 g tea bag that had to be prepared in a standard way for one week (washout period). Patients in the test group were instructed to have 300, 450, and 600 ml (2, 3, and 4 cups, respectively) in weeks 2, 3 and 4 respectively. We assessed the change in serum glutathion, superoxidismutase, total antioxidant capacity, FBS, CRP, HbA1C, lipid profiles and fibrinogen during the end of each week.

ELIGIBILITY:
Inclusion Criteria:

* Clinical diagnosis of type 2 diabetes mellitus

Exclusion Criteria:

* Intake of antioxidant supplements during previous six months

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 45 (Actual)
Dates: Start 2006-10; Primary Completion 2006-12 (Actual); Study Completion 2007-11 (Actual)

PRIMARY OUTCOMES:
Insulin Sensitivity, oxidative Stress, lipid Profile | 4 Weeks

CONTACTS AND LOCATIONS:
Overall Officials: Tirang R. Neyestani, Ph.D., Study Chair — National Nutrition & Food technology Research institute, Shaheed Beheshti University (M.C.), Islamic Republic of Iran,
Locations (1):
- National Nutrition and Food Technology Research Institute, Tehran, Tehran Province, Iran